CLINICAL TRIAL: NCT03536208
Title: Biological Effect of Warfarin on Pancreatic Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: no accrual for over 12 months
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Muhammad Beg, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 022018-090
Record Dates: First submitted 2018-03-28; First posted 2018-05-24 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Warfarin

STUDY DESIGN:
Intervention Model Description: patients will be assigned to warfarin by mouth daily on an outpatient basis. The first 5 patients enrolled will be assigned to the 1 mg QD dose level, the next 5 patients enrolled will be assigned to the 2 mg QD dose level, and so forth until all dose levels enrolled 5 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Warfarin (Experimental): Patients will be assigned to warfarin by mouth daily on an outpatient basis. Dose level will increase after 5 patients enrolled. Dose 1 = 1 mg warfarin; Dose 2 = 2 mg warfarin; Dose 3 = 2.5 mg warfarin; Dose 4 = 4 mg warfarin and Dose 5 = 5 mg warfarin
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — 5 different doses of warfarin will be assigned, ranging from 1mg to 5 mg.

SUMMARY:
This study aims to asses the effect of warfarin on markers of AXL pathway in patients with pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
There is emerging evidence from pre-clinical models that Axl activation is critical for the tumorigenesis and metastasis of pancreatic cancer. Warfarin is a readily available drug in the clinical setting and could be easily, safely, and quickly used in patients in combination with known cytotoxic chemotherapies to improve overall survival.

Oral warfarin has been well tolerated in both prophylaxis for catheter-associated thrombosis and in advanced pancreatic cancer patients.

The aim of this trial is to confirm the preclinical evidence that warfarin affects AXL pathway in patients with pancreatic cancer. This will validate the effect of escalating doses of warfarin on circulating biomarkers of AXL.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed, localized or metastatic adenocarcinoma of the pancreas. Diagnostic biopsy must be obtained at the study institution prior to enrollment. Pathology material must be available for review.
* Patient must have measurable disease per RECIST criteria
* Started most recent systemic therapy regimen within 15 days of enrollment (any line of therapy is allowed).
* Ability to tolerate, swallow and absorb oral medications.
* Ability to understand and the willingness to sign a written informed consent.
* Age > 18 years
* Negative blood pregnancy test within seven days of study entry for WOCBP
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

Exclusion Criteria:

* Active radiation therapy, or planned radiation therapy during study period
* Subjects may not be receiving any other investigational agents.
* Pregnant, nursing or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be potentially teratogenic.
* Underlying condition which may increase the risk of complications from warfarin therapy. These can include:

Known major bleeding diathesis:

* Coagulopathy
* Significant GI bleed within 6 months,
* Clinically significant hematuria or hemoptysis,
* Thrombolytic therapy within one month of study entry,
* Active peptic ulcer disease with bleeding. - Significant infection or other coexistent medical condition that would preclude protocol therapy including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Determine change in AXL pathway | 30 days
  Determine change in circulating biomarkers of AXL pathways (including phosphogas6, soluble AXL).

SECONDARY OUTCOMES:
Assess adverse events | 30 days
  Assess the adverse events (per CTCAE v4.0 criteria) associated with the addition of warfarin in patients with pancreatic cancer receiving chemotherapy.
Effect of warfarin on tissue markers | 30 days
  Evaluate the effect of warfarin on tissue markers of the AXL pathways measured by western blot analysis in tumor tissue and expression levels of EMY markers following warfarin therapy.
Antitumor effect | 30 days
  Antitumor effects will be observed by change in CA9-19 levels pre and post warfarin. therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad S Beg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States